CLINICAL TRIAL: NCT07261527
Title: Characterization of Skin and Facial Fat Pad Thickness Changes Following Microneedling Radiofrequency With and Without Topical Poly-L-Lactic Acid for Facial Rejuvenation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Ying Chen, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-25-0585
Record Dates: First submitted 2025-11-22; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Skin Texture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- microneedling radiofrequency (RF) (Experimental)
  Interventions: Device: microneedling RF treatment
- no treatment (No Intervention)
- microneedling RF treatment with topical poly-L-lactic acid (PLLA) (Experimental)
  Interventions: Device: microneedling RF treatment; Device: PLLA
- microneedling RF treatment with placebo (Experimental)
  Interventions: Device: microneedling RF treatment; Drug: Sterile Water as control

INTERVENTIONS:
Device: microneedling RF treatment — Participants will undergo two microneedling RF treatment sessions, 4-6 weeks apart
  Arms: microneedling RF treatment with placebo; microneedling RF treatment with topical poly-L-lactic acid (PLLA); microneedling radiofrequency (RF)
Device: PLLA — Participants will undergo two microneedling RF treatment sessions, 4-6 weeks apart followed by PLLA application after each treatment
  Arms: microneedling RF treatment with topical poly-L-lactic acid (PLLA)
Drug: Sterile Water as control — Participants will undergo two microneedling RF treatment sessions, 4-6 weeks apart followed by sterile water application after each treatment
  Arms: microneedling RF treatment with placebo

SUMMARY:
The purpose of this study is to evaluate whether microneedling RF subcutaneous fat pad thickness in the temple, submental, and cheek regions, to determine whether the addition of topical PLLA after microneedling RF alters or preserves subcutaneous fat pad thickness and to assess patient satisfaction and perceived outcomes following microneedling RF ± PLLA treatment.

ELIGIBILITY:
Inclusion Criteria:

* Seeking facial rejuvenation for cosmetic concerns
* Able and willing to provide informed consent
* Willing to comply with study procedures and follow-up visits

Exclusion Criteria:

* Prior filler injection or energy-based device treatment to the face within the past 6 months
* Previous facial surgeries
* Pregnant or breastfeeding
* Active infection, dermatitis, or open lesions in the treatment area
* History of keloids or abnormal scarring
* Known allergy to poly-L-lactic acid (PLLA)- Current participation in another clinical trial involving facial aesthetic treatments
* Presence of pre-cancerous or cancerous lesions in the treatment area
* Current or planned use of glucagon-like peptide-1 receptor agonists (e.g., Ozempic, semaglutide) during the study period. Subjects on these medications will be excluded due to potential effects on facial fat and overall weight.
* HIV+ patients
* Patients on HIV medications- Patients that have eczema and rosacea

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-24 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in subcutaneous fat pad thickness as measured by high-frequency ultrasound imaging | Baseline, 6 months

SECONDARY OUTCOMES:
Difference in fat pad thickness between the RF+PLLA side and RF-only side as assessed by ultrasound imaging | 6 months
Patient reported overall improvement in appearance as assessed by the Global Aesthetic Scale | 6 months
  This is scored on a 5 point scale from 1(much worse) to 5 (much improved) , higher score indicating better outcome
Change in satisfaction with forehead as assessed by the patient questionnaire | Baseline, 6 months
  This is scored from 1 (lowest) to 10 (highest)
Change in satisfaction with cheek as assessed by the patient questionnaire | Baseline, 6 months
  This is scored from 1 (lowest) to 9 (highest)
Change in satisfaction with submental as assessed by the patient questionnaire | Baseline, 6 months
  This is scored from 1 (lowest) to 9 (highest)
Change in overall social confidence as assessed by the patient questionnaire | Baseline, 6 months
  This is scored from 1 (lowest) to 10 (highest)

CONTACTS AND LOCATIONS:
Overall Officials: Ying Chen, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States